CLINICAL TRIAL: NCT01168596
Title: Rasagiline for the Symptomatic Treatment of Fatigue in Parkinson's Disease: A Bi-Center, Placebo-Controlled Study (The REST Fatigue Trial)
Brief Title: Rasagiline for the Symptomatic Treatment of Fatigue in Parkinson's Disease
Acronym: REST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20091035
Record Dates: First submitted 2010-02-19; First posted 2010-07-23 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator): Placebo tablet, 1 per day, duration is approximately 12 weeks.
  Interventions: Drug: Placebo
- rasagiline (Active Comparator): Rasagiline tablet, 1 mg, 1 per day, duration is approximately 12 weeks.
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — Comparison of Rasagiline versus placebo.
  Rasagiline tablet, 1 mg, 1 per day, duration is approximately 12 weeks.
  Other Names: Azilect
  Arms: rasagiline
Drug: Placebo — Comparison of Rasagiline versus placebo. Placebo tablet, 1 per day, duration is approximately 12 weeks.
  Arms: sugar pill

SUMMARY:
The purpose of the research study is to determine if rasagiline is an effective treatment for fatigue in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Despite the fact that fatigue affects 40-50% of all patients with PD and is a leading cause of disability, we currently do not have any effective treatments for this symptom. Rasagiline is a well-tolerated and effective treatment for the motor symptoms of PD. Rasagiline is a MAO-B inhibitor that may decrease the breakdown of dopamine. Many patients report an improvement in their energy levels when on this medication. A proven treatment for PD fatigue would significantly improve the quality of life for numerous patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of idiopathic PD by a movement disorders specialist. All subjects will be diagnosed using the UK Brain Bank criteria (Hughes et al., 1992).
2. Age between 40-85 years.
3. Able to sign and understand informed consent; and cognitively able to carry out the procedures in the study
4. Stable on all PD medications for at least 30 days; and psychotropic medications for at least 90 days.
5. Treatment naïve subjects who are appropriate candidates to begin MAO-inhibitor monotherapy as treatment for their PD may also be included in this study.
6. Fatigue Severity Scale ≥ 36 (KRupps et al., 1989)

Exclusion Criteria:

1. Clinically significant medical disease that is associated independently with fatigue (e.g. significant cardiac or pulmonary disease, anemia, obstructive sleep apnea, liver or kidney failure).
2. History of neurological illnesses other than PD or a history of a significant head trauma (involving unconsciousness).
3. Evidence of secondary or atypical parkinsonism as suggested by the presence of any of the following: 1) history of stroke(s), 2) exposure to toxins or neuroleptics, 3) history of encephalitis, 4) neurological signs of upper motor neuron disease, cerebellar involvement, supranuclear gaze palsy, or significant orthostatic hypotension.
4. MRI or CT scan with significant evidence of brain atrophy or other abnormalities (e.g. lacunar infarcts or iron deposits in the putamen.
5. Clinical diagnoses of dementia; or an MMSE score of < 25.
6. Unstable, newly diagnosed, or newly treated (i.e. less than 3 months) major psychiatric disorder such as depression or anxiety
7. Beck's Depression Inventory score >14.
8. Current or prior placement of Deep Brain Stimulator.
9. Currently taking an MAO-B inhibitor or medications which are used as fatigue treatments, including amantadine, modafinil, methylphenidate, atomoxetine or other psychostimulants.
10. Previously taken an MAO-B inhibitor for more than 2 weeks.
11. Hypersensitivity to rasagiline or its products
12. On mirtazapine, venlafaxine, regular use of compounds with vasoconstrictors, tramadol, meperidine, propoxyphene, dextromethorphan, St. John's wort, cyclobenzaprine
13. On omeprazole, ciprofloxacin or drugs that are metabolized through CYP1A2

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene A Malaty, MD, Principal Investigator — University of Florida Department of Neurology
Locations (3):
- United States (3):
  - University of Colorado Anschutz outpatient Pavilion, Aurora, Colorado
  - Shands and University of Florida Medical Plaza, Gainesville, Florida
  - Cleveland Clinic Center for Neurological Restoration, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Rasagiline: Rasagiline tablet, 1 mg, 1 per day, duration is approximately 12 weeks.
  Rasagiline : Comparison of Rasagiline versus placebo.
  Rasagiline tablet, 1 mg, 1 per day, duration is approximately 12 weeks.
- Sugar Pill: Placebo tablet, 1 per day, duration is approximately 12 weeks.
  Placebo : Comparison of Rasagiline versus placebo. Placebo tablet, 1 per day, duration is approximately 12 weeks.
Period: Overall Study
Arm/Group | Rasagiline | Sugar Pill
Started | 16 | 14
Completed | 13 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline | Sugar Pill | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.67 (7.39) | 65.43 (6.42) | 67.1 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: The MFIS rates how much of a problem fatigue has caused the subjects during the past month, including the day of testing. It consists of 21 questions of fatigue on quality of life. Each subject is asked to circle the appropriate response for each item: 0=never, 1=rarely, 2=sometimes, 3=often, 4=always, 5=almost always. The minimum score is 0 and the maximum is 105. The higher the score, the more fatigue the subject.
Time Frame: Change from baseline to week 12
Population: The number of patients used to calculate the results for this measure are different from the number of patients listed in the Participant Flow Module because of missing data. Any missing values were omitted from the summaries. Summary measures are for complete data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | 12.92 [.68 to 25.16] | 12.69 [1.4 to 23.98]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.81, Regression, Linear; Slope = 1.30, 95% CI 2-sided [-9.13 to 11.73], Standard Error of Mean 5.26

2. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Score consists of a nine-item questionnaire to identify common features of fatigue. Patients are instructed to choose a number from 1 to 7 that indicates their degree of agreement with each statement, where 1 = strongly disagree and 7 = strongly agree. Scores can range from a minimum of 9 to a maximum of 63. The higher the score, the more fatigue the subject.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 13
units on a scale | 12.38 [4.37 to 20.4] | 2.25 [-5.48 to 9.98]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.23, Regression, Linear; Slope = 4.38, 95% CI 2-sided [-2.75 to 11.51], Standard Error of Mean 3.60

3. Secondary Outcome: Multidimensional Fatigue Inventory (MFIS)
Description: The Multidimensional Fatigue Inventory (MFIS) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Subjects are instructed to choose a number from 1 to 5 that indicates their degree of agreement with each statement where 1 indicates that it is true and 5 that it is not true. There are positive and negative statements in the questionnaire. The range is 1 to 100, the higher the number the higher the fatigue.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 13
units on a scale | 2.62 [-4.15 to 9.38] | 6.83 [-0.02 to 13.69]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.75, Regression, Linear; Slope = 1.61, 95% CI 2-sided [-8.37 to 11.59], Standard Error of Mean 5.03

4. Secondary Outcome: PD Quality of Life Scale (PDQ39)
Description: PD Quality of Life Scale (PDQ39) is a 39-item questionnaire, which measures eight dimensions of health (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication and bodily discomfort) over the past 30 days. Dimension scores are coded on a scale of 0 (never) to 5 (always). The higher the score, the worse the quality of life affected by PD. The range for this test is 0 to 195. All eight dimensions are added for a total score.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | 7.54 [-1.61 to 16.69] | 5.67 [-1.87 to 13.21]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.54, Regression, Linear; Slope = 1.88, 95% CI 2-sided [-4.18 to 7.94], Standard Error of Mean 3.06

5. Secondary Outcome: Paced Auditory Serial Addition Test (PASAT)
Description: The Paced Auditory Serial Addition Test (PASAT) is a neuropsychological test used to assess capacity and rate of information processing and sustained and divided attention. Where subjects are given a number (every 3 seconds for the first series and 2 seconds for the second series) and are asked to add the number they just heard with the number they heard before. This is a challenging task that involves working memory, attention, and arithmetic capabilities.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -11.31 [-18.69 to -3.93] | -10.31 [-20.27 to -0.35]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.42, Regression, Linear; Slope = -5.17, 95% CI 2-sided [-17.76 to 7.43], Standard Error of Mean 6.36

6. Secondary Outcome: Finger Tapping
Description: The patient is asked to use the index finger on the side most affected by Parkinson's disease to tap for sixty seconds with the number of taps at 30 seconds and 60 seconds recorded.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: finger taps per sixty seconds
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
finger taps per sixty seconds | .46 [-.038 to 1.3] | -0.23 [-0.89 to .43]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.44, Regression, Linear; Slope = 0.36, 95% CI 2-sided [-0.56 to 1.29], Standard Error of Mean 0.47

7. Secondary Outcome: Hand-grip Strength
Description: The patients use the hand on the side most affected by Parkinson's disease to grip the dynamometer with as much strength as they can for 3 consecutive tries. The highest score will be their maximal voluntary contraction (MVC). The subject then rests for 60 seconds. The subject is asked to try to maintain 70% of their MVC and the duration the subject is able to maintain above 50% of their MVC is recorded. Immediately after the maintenance test, the subject performs three more MVCs and each one is recorded. These results are the duration the subject is able to maintain above 50% of their MVC.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
seconds | -9.08 [-23.86 to 5.69] | -8.36 [-17.42 to 0.7]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.82, Regression, Linear; Slope = 2.27, 95% CI 2-sided [-17.59 to 22.13], Standard Error of Mean 10.02

8. Other Pre Specified Outcome: Parkinson's Disease Sleep Scale (PDSS)
Description: The Parkinson's disease sleep scale (PDSS) is a 15-item visual analogue scale that assesses the profile of nocturnal disturbances in Parkinson's disease patients. The severity of symptoms of sleep over the past week is marked with a cross along a 10 cm line (labeled worst to best state). Responses are quantified by measuring the distance along each line to the intersection with the cross in centimetres, to the nearest 0.1 cm. The scores for each item range from 0 (symptom severe and always experienced) to 10 (symptom-free). The maximum score for PDSS is 150.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -13.46 [-24.04 to -2.88] | .64 [-9.1 to 10.38]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.52, Regression, Linear; Slope = -4.73, 95% CI 2-sided [-19.31 to 9.85], Standard Error of Mean 7.36

9. Other Pre Specified Outcome: Marin Apathy Inventory (Apathy Evaluation Scale)
Description: The Marin Apathy Inventory (Apathy Evaluation Scale) is a 14-item inventory measuring apathy of the subject over the past 2 to 4 weeks. Subjects are instructed to choose an answer from 0 to 3: 0=not at all, 1 = slightly, 2 = some, 3 = a lot, to questions related to apathy. The range would be 0 to 42, the higher the score the worse the apathy.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | .23 [-1.21 to 1.67] | .46 [-1.22 to 2.15]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.93, Regression, Linear; Slope = 0.11, 95% CI 2-sided [-2.15 to 2.36], Standard Error of Mean 1.14

10. Other Pre Specified Outcome: Visual Analog Scale - Subset: Afraid
Description: The Visual Analog Scale is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The severity of attitude at the time of testing is marked with a cross along a 10 cm line (labeled neutral to afraid, confused, sad, angry, energetic, tired, happy or tense). Responses are quantified by measuring the distance along each line to the intersection with the cross in centimetres, to the nearest 0.1 cm. The scores for each item range from 0 (symptoms-free) to 10 (symptom severe).
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -.77 [-2.08 to .55] | -.83 [-1.91 to .24]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.82, Regression, Linear; Slope = -0.11, 95% CI 2-sided [-1.05 to 0.83], Standard Error of Mean 0.47

11. Other Pre Specified Outcome: State-Trait Anxiety Inventory (STAI)
Description: The State-Trait Anxiety Inventory (STAI) is 40-item psychological inventory based on a 4-point Likert scale. Higher scores are positively correlated with higher levels of anxiety. The range for this test is 0 to 160.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | 3.62 [-7.37 to 14.6] | 6.08 [-5.56 to 17.72]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.56, Regression, Linear; Slope = -4.53, 95% CI 2-sided [-19.74 to 10.69], Standard Error of Mean 7.68

12. Other Pre Specified Outcome: Becks Depression Inventory (BDI-II)
Description: The Becks Depression Inventory (BDI-II) is a 21-question inventory measuring the severity of depression. Each subject is instructed to choose an answer on a scale value of 0 to 3 with the total score from 0 to 63. Higher total scores indicate more severe depressive symptoms.
Time Frame: Change from baseline to week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 16 | 14
units on a scale | 3.69 [-1.89 to 9.27] | 2.31 [.01 to 4.6]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.45, Regression, Linear; Slope = -2.21, 95% CI 2-sided [-8.02 to 3.59], Standard Error of Mean 2.93

13. Other Pre Specified Outcome: Unified Parkinson's Disease Rating Scale - Motor (UPDRS Part III)
Description: Unified Parkinson's Disease Rating Scale - Motor (UPDRS Part III)is a 14-question inventory measuring the motor functions of patients with Parkinson's Disease. Each subject is rated on a scale of 0 to 4 with the total score from 0 to 56. Higher total scores indicate more impairment of motor function.
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | 7.5 [0.6 to 14.4] | -0.83 [-4.71 to 3.04]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.58, Regression, Linear; Slope = 2.76, 95% CI 2-sided [-7.02 to 12.55], Standard Error of Mean 4.94

14. Other Pre Specified Outcome: Visual Analog Scale - Subset: Confused
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -.35 [-1.72 to 1.03] | -.21 [-1.39 to .98]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.95, Regression, Linear; Slope = 0.04, 95% CI 2-sided [-1.04 to 1.11], Standard Error of Mean 0.54

15. Other Pre Specified Outcome: Visual Analog Scale - Subset: Sad
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -.19 [-2.52 to 2.14] | -.5 [-1.82 to .82]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.48, Regression, Linear; Slope = -0.38, 95% CI 2-sided [-1.45 to 0.69], Standard Error of Mean 0.54

16. Other Pre Specified Outcome: Visual Analog Scale - Subset: Angry
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | .19 [-.81 to 1.2] | .33 [-0.55 to 1.21]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.84, Regression, Linear; Slope = -0.07, 95% CI 2-sided [-0.71 to 0.58], Standard Error of Mean 0.33

17. Other Pre Specified Outcome: Visual Analog Scale - Subset: Energetic
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | -1.19 [-3.27 to .88] | -2.12 [-4.33 to 0.08]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.44, Regression, Linear; Slope = 0.49, 95% CI 2-sided [-0.77 to 1.76], Standard Error of Mean 0.64

18. Other Pre Specified Outcome: Visual Analog Scale - Subset: Tired
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | .04 [-2.59 to 2.67] | .75 [-1.32 to 2.82]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.71, Regression, Linear; Slope = -0.33, 95% CI 2-sided [-2.06 to 1.41], Standard Error of Mean 0.88

19. Other Pre Specified Outcome: Visual Analog Scale - Subset: Happy
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 15 | 14
units on a scale | .04 [-3.14 to 3.22] | -0.33 [-2.77 to 2.10]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.31, Regression, Linear; Slope = 0.64, 95% CI 2-sided [-0.62 to 1.90], Standard Error of Mean 0.64

20. Other Pre Specified Outcome: Visual Analog Scale - Subset: Tense
Description: as for outcome 10
Time Frame: Change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Sugar Pill
Number analyzed (Participants) | 14 | 14
units on a scale | .25 [-1.02 to 1.52] | .83 [-0.47 to 2.13]
Statistical Analysis 1: Comparison: Rasagiline vs Sugar Pill; Test type: Superiority or Other; p = 0.94, Regression, Linear; Slope = -0.06, 95% CI 2-sided [-1.68 to 1.56], Standard Error of Mean 0.82

ADVERSE EVENTS:
Arm/Group | Rasagiline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/14
Other Adverse Events (participants affected / at risk) | 9/16 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=16) | Sugar Pill (N=14)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) — Thought by PI to be unlikely related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=16) | Sugar Pill (N=14)
exostosis foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — bone spur on left foot. Moderate in severity. Thought by the PI to be unrelated to the study.
dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Intermittent dizzy spells reported by patient. PI thought it unlikely to be related to study medication.
Headache (Nervous system disorders) | 1 (1) | 2 (3) — Patient reported having headaches occasionally in the past but now having worsened headache meaning the pain was slightly worse when he had headaches. The PI thought it unlikely to be related to the study medication.
depression (Psychiatric disorders) | 1 (1) | 1 (1) — Patient on active drug had depression already and reported a worsening of depression symptoms. PI thought to be unrelated to the study medication. Sub-I felt patient on placebo was unlikely related to study medication.
insomnia (Psychiatric disorders) | 1 (1) | 0 (0) — PI thought it unlikely to be related to the study medication.
hypertension (Vascular disorders) | 0 (0) | 1 (1)
thrombolembolic event (Vascular disorders) | 1 (1) | 0 (0) — blood clot in left calf reported by patient. Thought by sub-I to be unrelated.
skin infection (Infections and infestations) | 1 (1) | 0 (0) — infection on left arm. Thought by sub-I to be unrelated to study medication.
urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient reported worsened urinary urgency. Thought by PI to be unrelated to study medication.
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Thought to be possibly related to study drug by sub-I.
urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) — PI and sub-I each thought their patient's UTI was unlikely related to the study medication.
nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) — The sub-I thought the 2 instances in one of the patients affected was possibly related to the study medication and the other patient's nausea was probably related to the study medication.
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Thought by PI to be unrelated to study medication.
upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) — Sub-I thought it unlikely hese were related to the study medication.
fatigue (General disorders) | 1 (1) | 1 (1) — Two patients reported worsened/increased fatigue which was thought by sub-I and PI unlikely to be related to study medication.
Fever (General disorders) | 1 (1) | 0 (0) — Patient reported fever only in the evening. PI thought it unlikely to be related to study medication.
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Body aches considered unlikely to be related to study medication by sub-I.
paresthesia (Nervous system disorders) | 0 (0) | 1 (1) — patient reported mild numbness in fingers - bilateral. Sub-I thought to be possibly related to study medication.
gait disturbance (General disorders) | 1 (1) | 0 (0) — Patient reported increased freezing. Thought to be unrelated to study medication by the PI.
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient reported right hip pain. Thought by PI to be unlikely related to study medication.
Gastrointestinal disorders - other, diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Diverticulitis thought by sub-I to be unlikely related to study medication.
Neoplasms benign, malignant and unspecified, other - squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — patient had a squamous cell carcinoma removed from right hand. Though by PI to be unrelated to study medication.
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient reported muscle cramp in right leg. Sub-I thought to be possibly related to study medication.
injury, poisoning and procedureal complications, other - skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — patient reported a skin tear (from tape) on left arm. Sub-I thought to be unrelated to study medication.
extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) — patient reported dyskinesias. Thought by PI to be possibly related to study medication.
urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient reported burning upon urination. PI thought it to be unrelated to study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No